CLINICAL TRIAL: NCT04140292
Title: Vitamin D Supplementation as a Neoadjuvant for Photodynamic Therapy of Actinic Keratoses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5619; NCT04482322 (obsolete NCT alias)
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Results first posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Study group will be compared to a baseline cohort of patients from a previous study (IRB 16-1615) who received the same regimen of PDT, but without any Vit D
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vitamin D3 + Photodynamic therapy (PDT) (Experimental): Patients receive Vitamin D3 10,000 IU daily for 5 or 14 days depending on VitD baseline level. They then undergo Photodynamic therapy (PDT) for treatment of actinic keratosis.
  Interventions: Drug: Photodynamic therapy (PDT); Drug: Vitamin D3

INTERVENTIONS:
Drug: Photodynamic therapy (PDT) — PDT is a technique that combines a photosensitizing drug and an intense light source to kill tumor cells
  Noninvasive fluorescence dosimetry may be performed on up to 6 lesions. Levulan Kerastick will be applied to each lesion and left to incubate for 30 minutes. Blue light (Blu-U device, 20 J/cm2, 33 minutes) will be administered.
Drug: Vitamin D3 — D3 pills (10,000 IU each) to be taken daily at home, beginning at either day -5 or day -14, as per their assignment
  Participants will receive a 5-day or 14-day supplementation of Vitamin D10,000 IU depending on their baseline Vitamin D 25 Hydroxy result

SUMMARY:
This study is open to individuals with Actinic Keratoses (skin lesions that have the potential to turn into skin cancer), who are receiving photodynamic therapy (PDT) as part of their clinical care. The purpose of this study is to test and demonstrate that vitamin D pre-treatment can enhance PDT efficacy in the treatment of Actinic Keratoses.

Participants will be asked to take vitamin D supplements prior to their standard of care PDT treatment.

Participation in the research will last about 3-4 months.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether acute supplementation (neoadjuvant Vitamin D3), adjusted according to baseline Vitamin D status, can improve the clinical PDT response relative to participants receiving PDT alone

The secondary objective of this study is to determine whether gene polymorphisms in VDR and CYP27B1 are predictive for the degree of responsiveness to Vitamin D as a neoadjuvant for PDT.

This study is a non-randomized interventional trial, in which the study group will be compared to a baseline cohort of patients from a previous study who received the same regimen of PDT, but without any Vit D. It is anticipated that 30 participants will be involved in this study.

ELIGIBILITY:
Inclusion Criteria:

* Actinic keratoses in sufficient numbers (>10) to warrant PDT therapy in the clinic
* Able to understand and willing to sign a written informed consent document
* Female subjects must not become pregnant during the study:

  * The effects of 5-aminolevulinic acid (LevulanTM) on the human fetus are unknown. For this reason, women of child-bearing potential must agree to use contraception (double barrier method of birth control or abstinence) prior to study entry, and throughout study participation. Should a woman become pregnant or suspect that she is pregnant while she is participating in this study, she should inform the treating physician immediately.

Exclusion Criteria:

* Pregnant or nursing.
* At risk for hypercalcemia (renal disease, sarcoidosis, etc.)
* Using topical retinoids, since these can exacerbate the post-PDT erythema reaction.
* Using any topical treatment on their AKs; must stop at least one month prior.
* Currently undergoing treatment for other cancers with medical or radiation therapy.
* Patients with a known hypersensitivity to 5-aminolevulinic acid or any component of the study material.
* Patients with history of a photosensitivity disease, such as porphyria cutanea tarda.
* Currently participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward V Maytin, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication

REFERENCES:
- [Derived] Bullock TA, Negrey J, Hu B, Warren CB, Hasan T, Maytin EV. Significant improvement of facial actinic keratoses after blue light photodynamic therapy with oral vitamin D pretreatment: An interventional cohort-controlled trial. J Am Acad Dermatol. 2022 Jul;87(1):80-86. doi: 10.1016/j.jaad.2022.02.067. Epub 2022 Mar 18. PMID 35314199

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D3 + Photodynamic Therapy (PDT): Patients receive Vitamin D3 10,000 IU daily for 5 or 14 days depending on VitD baseline level. They then undergo Photodynamic therapy (PDT) for treatment of actinic keratosis.
  Photodynamic therapy (PDT): PDT is a technique that combines a photosensitizing drug and an intense light source to kill tumor cells
  Noninvasive fluorescence dosimetry may be performed on up to 6 lesions. Levulan Kerastick will be applied to each lesion and left to incubate for 30 minutes. Blue light (Blu-U device, 20 J/cm2, 33 minutes) will be administered.
  Vitamin D3: D3 pills (10,000 IU each) to be taken daily at home, beginning at either day -5 or day -14, as per their assignment
  Participants will receive a 5-day or 14-day supplementation of Vitamin D10,000 IU depending on their baseline Vitamin D 25 Hydroxy result
- Photodynamic Therapy (PDT): Participants will be matched to other participants from a prior study (NCT03467789) involving PDT only, based on their baseline vitamin D level. These participants were used as a control group.
Period: Overall Study
Arm/Group | Vitamin D3 + Photodynamic Therapy (PDT) | Photodynamic Therapy (PDT)
Started | 33 | 42
Completed | 29 | 26
Not Completed | 4 | 16
Not completed — Restriction on outpatient visits due to COVID-19. | 4 | 16

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Photodynamic Therapy (PDT): Data for the participants in this arm are from a previous basic science study that looked at Vit D level that got standard of care PDT. These participants were used as a control group.
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 + Photodynamic Therapy (PDT) | Photodynamic Therapy (PDT) | Total
Number analyzed (Participants) | 29 | 26 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 17 | 13 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 27 | 23 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 29 | 26 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 26 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical PDT Response as Measured by Percent Change in AK Lesions From Baseline to 3 Months
Description: Clinical PDT response as measured by the percent change of AK lesions 3 months after treatment
  Baseline vitamin D (calcidiol) level will be taken for each patient.
Time Frame: 3 months after treatment
Population: Participants who received treatment.
Measure: Mean (Standard Deviation); unit: Percent change of AK lesions
Arm/Group | Vitamin D3 + Photodynamic Therapy (PDT) | Photodynamic Therapy (PDT)
Number analyzed (Participants) | 29 | 26
Percent change of AK lesions | 59.1 (15.9) | 72.5 (13.6)

2. Secondary Outcome: Correlation Between Vitamin D Receptor (VDR) Polymorphisms and Percent Reduction in AK
Description: Whether gene polymorphisms in VDR and CYP27B1 are predictive for the degree of responsiveness (as measured by percent reduction in AK) to Vitamin D as a neoadjuvant for PDT.
Time Frame: 3 months after treatment
Population: Unable to obtain any information about the PpIX accumulation levels because fluorescence imaging dosimeter broke down and it was unable to be replaced.
Arm/Group | Vitamin D3 + Photodynamic Therapy (PDT) | Photodynamic Therapy (PDT)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Reporting 1 or Higher on the Pain Scale
Description: Pain scale recorded on a 0-to-10 visual/analog scale, with higher scores mean more pain; 0 is no pain, 10 is "the worst pain imaginable". Number of participants receiving treatment that reported a pain level greater than 1.
Time Frame: During treatment (at the 5 min mark), and again immediately afterwards.
Population: Participants that received treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Vitamin D3 + Photodynamic Therapy (PDT): Participants receive Vitamin D3 10,000 IU daily for 5 or 14 days depending on VitD baseline level. They then undergo Photodynamic therapy (PDT) for treatment of actinic keratosis.
  Photodynamic therapy (PDT): PDT is a technique that combines a photosensitizing drug and an intense light source to kill tumor cells
  Noninvasive fluorescence dosimetry may be performed on up to 6 lesions. Levulan Kerastick will be applied to each lesion and left to incubate for 30 minutes. Blue light (Blu-U device, 20 J/cm2, 33 minutes) will be administered.
  Vitamin D3: D3 pills (10,000 IU each) to be taken daily at home, beginning at either day -5 or day -14, as per their assignment
  Participants will receive a 5-day or 14-day supplementation of Vitamin D10,000 IU depending on their baseline Vitamin D 25 Hydroxy result
Arm/Group | Vitamin D3 + Photodynamic Therapy (PDT) | Photodynamic Therapy (PDT)
Number analyzed (Participants) | 29 | 26
Participants | 0 | 0

4. Secondary Outcome: Tolerability as Measured by Participants' Symptom Score Sheets
Description: Participants are asked to recall the symptoms they experienced during the week following PDT. The study physician asks them whether they had experienced each of the following 13 symptoms (YES/NO), and positive (YES) answers were summed to create a Side Effects Score (SES). The maximum and minimum possible values are 13 and 0 respectively, with a higher score correlating to poorer participant outcomes.
  The 13 possible side effects were: pain, erythema, scabbing, blistering, erosions, edema, warmth, exfoliation, discharge, hemorrhage, tightness, hyperpigmentation, hypopigmentation.
Time Frame: 1 week after treatment
Population: Participants who received treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin D3 + Photodynamic Therapy (PDT) | Photodynamic Therapy (PDT)
Number analyzed (Participants) | 29 | 26
score on a scale | 3.7 (2.2) | 3.7 (1.9)

5. Secondary Outcome: Accumulation of Protoporphyrin IX (PpIX) Within AK
Description: Accumulation of protoporphyrin IX (PpIX) within AK
  PpIX accumulation in areas of both actinic damage and normal skin will be measured with a fluorescence dosimeter. The level of calcidiol, a clinically accepted marker of vitamin D status, will be measured in each patient to see if supplementation with 10,000 IU of Vitamin D increase the accumulation
Time Frame: 3 months after treatment
Population: as for outcome 2
Arm/Group | Vitamin D3 + Photodynamic Therapy (PDT) | Photodynamic Therapy (PDT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No AE or SAEs were collected.
Description: No AE or SAEs were collected.
Arm/Group | Vitamin D3 + Photodynamic Therapy (PDT) | Photodynamic Therapy (PDT)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT04140292/Prot_SAP_002.pdf
  • Informed Consent Form (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT04140292/ICF_003.pdf